CLINICAL TRIAL: NCT00116207
Title: Oxidative Stress and Cardiovascular Denervation in Diabetes: An Interventional Trial
Brief Title: An Intervention Trial for Cardiac Neuropathy in Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Rodica Pop-Busui, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB:2002-0460
Record Dates: First submitted 2005-06-27; First posted 2005-06-28 (Estimated); Results first posted 2016-01-05 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-06

CONDITIONS: Diabetic Autonomic Neuropathy
Keywords: Type 1 Diabetes; Oxidative Stress; Diabetic Complications; Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus, Type 1; Diabetes Complications | interventions — Antioxidants; Allopurinol; Niacinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ORAL ANTIOXIDANT (Experimental): Allopurinol (300mg daily), ALA (600mg twice daily) nicotinamide (750 mg twice daily) Given orally These drugs were given together as a combination and not as individual treatment.
  Interventions: Drug: ORAL ANTIOXIDANT
- Placebo (Placebo Comparator): Placebo administered twice daily.
  Interventions: Drug: ORAL ANTIOXIDANT

INTERVENTIONS:
Drug: ORAL ANTIOXIDANT — Comparison of triple antioxidant combination therapy vs placebo.
  Other Names: Allopurinol (300mg daily),; ALA (600mg twice daily); nicotinamide (750 mg twice daily)

SUMMARY:
The focus of this project is cardiovascular diabetic autonomic neuropathy (DAN). DAN affects the nerves that control heart rate and blood flow to the heart in people with diabetes. DAN may cause problems with the rhythm of the heartbeat or decrease blood flow to the heart. Three medications will be tested for their effectiveness in DAN.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* A1C <9%
* Mild neuropathy
* Mild retinopathy
* Mild nephropathy

Exclusion Criteria:

* History of drug or alcohol dependence, heart disease, viral illness, liver disease, advanced kidney disease
* Pregnant or nursing
* Severely overweight

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2000-01; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva L Feldman, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pop-Busui R, Stevens MJ, Raffel DM, White EA, Mehta M, Plunkett CD, Brown MB, Feldman EL. Effects of triple antioxidant therapy on measures of cardiovascular autonomic neuropathy and on myocardial blood flow in type 1 diabetes: a randomised controlled trial. Diabetologia. 2013 Aug;56(8):1835-44. doi: 10.1007/s00125-013-2942-9. Epub 2013 Jun 6. PMID 23740194

RESULTS

PARTICIPANT FLOW:
Groups:
- ORAL ANTIOXIDANT: Allopurinol (300mg daily), ALA (600mg twice daily) nicotinamide (750 mg twice daily) Given orally
  ORAL ANTIOXIDANT: Comparison of triple antioxidant therapy to placebo
- Placebo: Placebo administered twice daily.
  ORAL ANTIOXIDANT: Comparison of triple antioxidant therapy to placebo
Period: Overall Study
Arm/Group | ORAL ANTIOXIDANT | Placebo
Started | 22 | 22
Completed | 13 | 18
Not Completed | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ORAL ANTIOXIDANT | Placebo | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (12) | 47 (10) | 46 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 13 | 18 | 31
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Global [11C]HED Retention Index (RI)
Description: Distal defects in [11C]meta-hydroxyephedrine ([11C]HED) retention involving at least 10 % of the left ventricle was used to define Cardiac Autonomic Neuropathy (CAN). The retention index (RI) is the unit of measure and is expressed as [11C]HEDblood min -1[ml tissue]-1
  PET Data of Randomized Subjects at Baseline and 24-Months
  The primary outcome was the change in the global [11C]HED RI = measure of cardiac innervation at 24 months in participants taking the active drug compared with those on placebo.
Time Frame: Baseline, 24 months
Measure: Mean (Standard Deviation); unit: Retention index
Arm/Group | ORAL ANTIOXIDANT | Placebo
Number analyzed (Participants) | 13 | 18
Retention index
  BASELINE | 0.081 (0.017) | 0.073 (0.016)
  24 MONTHS | 0.070 (0.018) | 0.074 (0.016)
Statistical Analysis 1: Comparison: ORAL ANTIOXIDANT vs Placebo; BASELINE; Test type: Superiority or Other; p = 0.32, ANOVA — p values were computed using a general linear model (ANOVA) adjusted at baseline for age, sex, HbA1c
Statistical Analysis 2: Comparison: ORAL ANTIOXIDANT vs Placebo; 24-MONTH; Test type: Superiority or Other; p = 0.045, ANOVA — p values were computed using a general linear model (ANOVA) adjusted at baseline for age, sex, HbA1c

2. Secondary Outcome: Global Coronary Flow Reserve as a Measure of Endothelial Function
Description: global myocardial blood flow reserve as a measure of endothelial function. Measured by PET using [13N]ammonia at rest and during adenosine stimulated coronary vasodilation.
Time Frame: Baseline, 24 months
Measure: Mean (Standard Deviation); unit: ratio (rest:stress)
Arm/Group | ORAL ANTIOXIDANT | Placebo
Number analyzed (Participants) | 13 | 18
ratio (rest:stress)
  BASELINE | 2.95 (1.32) | 2.94 (1.70)
  24 MONTH | 3.02 (1.82) | 3.22 (0.85)
Statistical Analysis 1: Comparison: ORAL ANTIOXIDANT vs Placebo; BASELINE; Test type: Superiority or Other; p = 0.52, ANOVA — p values were computed using a general linear model (ANOVA) adjusted at baseline for age, sex, HbA1c
Statistical Analysis 2: Comparison: ORAL ANTIOXIDANT vs Placebo; 24 MONTH; Test type: Superiority or Other; p = 0.82, ANOVA — p values were computed using a general linear model (ANOVA) adjusted at baseline for age, sex, HbA1c

3. Secondary Outcome: Systemic Oxidative Stress
Description: ng of 8-epi prostaglandin F2alpha /G creatinine assessed in 24 hour urine collection
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: ng/G creatinine
Arm/Group | ORAL ANTIOXIDANT | Placebo
Number analyzed (Participants) | 13 | 18
ng/G creatinine | 2.92 (1.99) | 2.09 (1.12)
Statistical Analysis 1: Comparison: ORAL ANTIOXIDANT vs Placebo; 24 MONTH; Test type: Superiority or Other; p = 0.24, ANOVA — p values were computed using a general linear model adjusted at baseline for age, sex, HbA1c

4. Secondary Outcome: Inflammation
Description: High Sensitivity CRP (nmol/L)
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | ORAL ANTIOXIDANT | Placebo
Number analyzed (Participants) | 13 | 18
nmol/L | 17.51 (20.19) | 16.95 (18.38)
Statistical Analysis 1: Comparison: ORAL ANTIOXIDANT vs Placebo; 24 MONTH; Test type: Superiority or Other; p = 0.83, ANOVA — p values were computed using a general linear model (ANOVA) adjusted at baseline for age, sex, HbA1c

ADVERSE EVENTS:
Time Frame: At each subject visit adverse events were reviewed with the subject.
Arm/Group | ORAL ANTIOXIDANT | Placebo
Serious Adverse Events (participants affected / at risk) | 1/22 | 1/22
Other Adverse Events (participants affected / at risk) | 18/22 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ORAL ANTIOXIDANT (N=22) | Placebo (N=22)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Liver cancer resulting in death
Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ORAL ANTIOXIDANT (N=22) | Placebo (N=22)
Non-Serious Adverse Events (General disorders) | 18 (137) | 21 (141) — General complaints or concerns reported by participants that were non-serious, and mild to moderate in nature

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No